CLINICAL TRIAL: NCT04075981
Title: Prevention of Post-operative Atrial Fibrillation by BOTulinum Toxin Injections Into Epicardial Fat Pads Around Pulmonary Veins in Patients Undergoing Cardiac Surgery"
Brief Title: Prevention Atrial Fibrillation by BOTulinum Toxin Injections (BOTAF)
Acronym: BOTAF
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Merz Pharmaceuticals (Industry); Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P170912J; PHRCN-17-0371 (Other: Ministry of health)
Record Dates: First submitted 2019-08-19; First posted 2019-09-03 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Cardiac Surgery
Keywords: Xeomin®; Botox; Botulinum; Atrial Fibrillation; Cardiac surgery
MeSH Terms: conditions — Atrial Fibrillation | interventions — Botulinum Toxins, Type A; incobotulinumtoxinA

STUDY DESIGN:
Intervention Model Description: The study is a double-blind multicenter randomized trial comparing treatment with botulinum toxin to normal saline (placebo) on top of usual treatment to prevent atrial fibrillation in patients undergoing cardiac surgery (coronary artery bypass graft surgery (CABG), aortic valve surgery, or ascending aorta surgery).
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Botulinum toxin (Experimental): All patients from the experimental group will receive botulinum toxin (Xeomin®, incobotulinumtoxin A, Merz Pharma GmbH & Co KGaA, Germany; 200 U dissolved in 4 mL of 0.9% normal saline and 50 U/1 mL will be injected at each fat pad).
  Botulinum toxin will be injected into the entire visible area of the 4 major epicardial fat pads, during extra corporal circulation and before aortic cross clamping in order to reduce the time of ischemia.
  The whole estimated dosage would be therefore 200 units of incobotulinumtoxin A,
  Interventions: Drug: Botulinum Toxin Type A Injection [Xeomin]
- Placebo (Placebo Comparator): All patients from the control group will receive placebo. Before the main stage of the surgery, during extra corporal circulation and before aortic cross clamping, the placebo dissolved in 4 mL of 0.9% normal saline will be injected into the entire visible area of the 4 major epicardial fat pads as follows (1 mL at each fat pad).
  Interventions: Other: Drug placebo

INTERVENTIONS:
Drug: Botulinum Toxin Type A Injection [Xeomin] — Before the main stage of the surgery, botulinum toxin will be injected into the entire visible area of the 4 major epicardial fat pads, during extra corporal circulation and before aortic cross clamping in order to reduce the time of ischemia.
  Other Names: Xeomin
  Arms: Botulinum toxin
Other: Drug placebo — All patients from the control group will receive placebo. Before the main stage of the surgery, during extra corporal circulation and before aortic cross clamping, the placebo will be injected into the entire visible area of the 4 major epicardial fat pads as follows (1 mL at each fat pad).
  Arms: Placebo

SUMMARY:
Over the past few years, research has focused on the prevention of atrial fibrillation (AF) after cardiac surgery, but highly effective interventions are still missing. Postoperative AF remains the most common complication after cardiac surgery, with an incidence of 10 to 50%. This complication is usually a transient condition that resolves spontaneously but it has major adverse consequences for patients and the health care system, including increased rates of death, complications (strokes), and hospitalisations with inflated costs.

Recently, animal studies have demonstrated that neurotoxins such as botulinum toxin (BTX) injected into fat pads could suppress AF inducibility by parasympathetic activation. Botulinum toxin injection in fat pads has been studied in the dog's heart and could be associated with the reduction of atrial fibrillation in postoperative cardiac surgery. One pilot study has demonstrated the feasibility and safety of this technique in the human heart.

The investigators hypothesize that botulinum toxin injection may substantially reduce postoperative AF during the first postoperative month after cardiac surgery without any serious adverse events. By the suppression of ganglionic plexi (GP) activity in the epicardial fat pads, mild term antiarrhythmic effects can be achieved with fewer antiarrhythmic drugs and anticoagulant treatment.

DETAILED DESCRIPTION:
Botulinium toxin use has been developed with success in wide-ranging fields (neurology, otorhinolaryngology, gynaecology, urology, plastic surgery, pain therapy), but not in cardiology.

In the cardio-vascular field, only one pilot study on man has shown its utility in the prevention of atrial fibrillation by blocking the triggering through the sympathic and parasympathic systems. The investigators need to assess its potential benefits to prevent postoperative atrial tachyarrhythmia in a randomised multicentre study, with an expected impact of approximately 30,000 patients per years in France undergoing these types of cardiac surgery.

The investigators hypothesize that botulinum toxin injection may substantially reduce postoperative AF during the first 3 weeks after cardiac surgery without any serious adverse events. By the suppression of ganglionic plexi (GP) activity in the epicardial fat pads, mild term antiarrhythmic effects can be achieved with fewer antiarrhythmic drugs and anticoagulant treatment.

ELIGIBILITY:
Inclusion Criteria:

* Indication for cardiac surgery (CABG, aortic valve repair or aortic valve replacement excluding the sutureless valve, ascending aorta surgery), according to the European Heart Association guidelines.
* Patients in hemodynamically stable condition.
* Sinus rhythm at moment of randomisation (ECG).
* Age: ≥18 to ≤80 years old.
* Negative serum or urinary β-hCG for women of child-bearing potential.
* Patients able to attend several consultations at the centre.
* Informed consent signed.
* Affiliation to French social security regime.

Exclusion Criteria:

* Previous cardiac surgery.
* Persistent AF or atrial tachycardia.
* Planned maze procedure or pulmonary vein (PV) isolation.
* Use of class I or III antiarrhythmic drugs within 5 elimination half-life of the drug (for amiodarone: one year).
* Mitral or tricuspid valve surgery.
* Congenital cardiomyopathy.
* Neuro-muscular disease (including disorders of pre-operative swallowing).
* Protected populations e.g. minor patient, breastfeeding women, patients under legal guardianship, curatorship or legal protection. .
* Participation in another interventional trial.
* Unwillingness to participate.
* Contraindications to botulinum toxin under investigation or to the excipients: known hypersensitivity.
* Patient with active endocarditis Minimal invasive surgery (ministernotomy)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants presenting at least one episode of atrial fibrillation (more than 30 seconds), during the first 3 weeks after cardiac surgery | 3 weeks
  An episode of AF will be considered part of the primary outcome analyses if it last at least 30 seconds continuously within 21 days after cardiac surgery and is documented by any form of monitoring, regardless of symptoms. The definition of atrial fibrillation (at least 30 seconds continuously) results from recent publications and AF definition in the cardiovascular field64.
  This endpoint will be measured through both holter ECG Spiderflash-t recorder during the first 21 days post-op and ECG daily monitoring during the first 7 days after surgery.

SECONDARY OUTCOMES:
Death rate | 12 months
  Death rate at 12 months
Number of participants presenting at least one episode of atrial fibrillation (more than 30 seconds), during the first 3 monthes after cardiac surgery | 3 months
  Incidence of rhythm disorders of postoperative AF in patients undergoing cardiac surgery at 3 months defined as atrial arrhythmia during at least 30 seconds continuously.
Number of patients presenting a cardiovascular event as conduction troubles, congestive heart failure, major bleeding, stroke, and arterial thromboembolic events | 3 months
  conduction troubles such as atrioventricular block or the need for transient or permanent placement of a pacemaker, congestive heart failure, major bleeding, stroke, and arterial thromboembolic events.cardiac surgery at 3 months defined as atrial arrhythmia during at least 30 seconds continuously.
Incidence of atrial tachyarrhythmia / Flutter | 3 months
  Incidence of all atrial tachyarrhythmia including atrial fibrillation, but also atrial flutter and atrial tachycardia 3 months, and each arrhythmia taken individually between the two parallel groups.cardiac surgery at 3 months defined as atrial arrhythmia during at least 30 seconds continuously.
New onset of postoperative AF | 3 months
  Incidence of new onset of postoperative AF depending on the following subgroups: age, gender, heart failure, left atrial enlargement, Euro SCORE 2, renal function, type of surgery
End of surgery until discharge (intervals from end of surgery to extubation, in hours) | 10 days
  Mechanical ventilation duration and postoperative length of stay in intensive care unit and in hospital
Readmission rate | 3 and 12 months
  Unplanned readmission rate at 3 months and 12 months for cardiovascular cause or haemorrhage.
Antiarrhythmic drugs | 3 months
  Number of antiarrhythmic drugs and curative anticoagulation within 3 months following cardiac surgery.
total hospital cost | twelve months
  Initial admission and readmissions for cardiovascular cause, and Incremental cost effectiveness ratio (additional cost per additional survival, additional QALY or per additional adverse event recognised).

CONTACTS AND LOCATIONS:
Overall Officials: FLORENS Emmanuelle, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (9):
- France (9):
  - Corentin Celton, Issy-les-Moulineaux, France
  - Hôpital Marie Lannelongue, Le Plessis-Robinson, France
  - CHU Limoges, Limoges, France
  - Hôpital Saint-Joseph, Marseille, Provence-Alpes-Côte d'Azur Region
  - Clinique Ambroise Paré, Neuilly-sur-Seine, Île-de-France Region
  - Institut Mutualiste Montsouris, Paris, Île-de-France Region
  - Hôpital Européen Georges Pompidou, Paris, Île-de-France Region
  - Hôpital Bichat, Paris, Île-de-France Region
  - Centre Cardiologique du Nord, Saint-Denis, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Yes
Individuel participant data that underlie results in publication could be shared Individuel participant data detailed in meta analysis protocol could be shared
Supporting Information: Study Protocol, ICF
Time Frame: one year after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on scientific project and scientific involvement of the PI team.
  Teams wishing obtain IPD must meet the sponsor and IP team to present scientifics (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization